CLINICAL TRIAL: NCT03916926
Title: Reducing Oral Health Disparities of Older Adults: Comparative Effectiveness of 2 Treatments
Brief Title: Older Adult Effectiveness of 2 Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Suchitra Nelson, Professor and Interim Chair, Department of Community Dentistry, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AD-2018-C1-10590
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Dental Caries
Keywords: Dental Caries; Oral Health Quality of Life
MeSH Terms: conditions — Dental Caries | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Intervention Model Description: The comparative effectiveness of "simple medical", i.e. SDF versus "typical dental", i.e. atraumatic restorative treatment (ART) + fluoride varnish (FV) intervention in this study is focused on the person level to address the unique oral health needs of low-income older adults.
  The interventions proposed for this study are in current clinical use. Both coronal and root surface tooth decay lesions will be treated. The two evidence-based strategies in older adults will be compared as follows:
  Arm 1 (N=295 participants): A "simple medical strategy" consisting of SDF versus Arm 2 (N=295 participants): A "typical dental strategy" consisting of ART + FV
Who Masked: Participant
Masking Description: We will attempt blinding of participants to the study group (participants). The hygienists (care providers) will be unaware of the treatment assignment when they go to their respective housing facilities. For all treatment visits, assessments will be conducted prior to the intervention delivery.
  Two hygienists will go to the housing facility randomized to the SDF arm and the other two will go to the ART + FV arm. The baseline treatment to be applied will be revealed only after the baseline caries exam has been completed. At the 6 month follow-up visit, the two hygienists that applied SDF will now go to the facilities randomized to the ART + FV facilities and vice-versa to conduct the 6-month follow up caries assessment exam and treatment. We will follow similarly for the 12-moth follow-up visit. By this strategy, we will make sure that potential bias of the hygienist evaluating their own work is minimized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- A "simple medical strategy" consisting of SDF (Experimental): The treatment will be bi-annual application (at baseline and 26 weeks) of topical 38% silver diamine fluoride (Advantage Arrest, Elevate Oral Care LLC., West Palm Beach, FL) following manufacturer's instructions and guidelines published by UCSF (2016).
  Interventions: Device: A "simple medical strategy" consisting of silver diamine fluoride (SDF)
- A "typical dental strategy" consisting of ART + FV (Active Comparator): Atraumatic Restorative Treatment (ART) will be a modification of the approach used by Lo and colleagues (2006), and the cavity restored at baseline with resin reinforced glass-ionomer cement (GIC) (GC Corporation, Japan). Participants in this arm will also receive biannual topical fluoride varnish application (FluoriMax, Elevate) according to manufacturer's instructions.
  Interventions: Device: B "typical dental strategy" consisting of atraumatic restorative treatment (ART) with glass ionomer cement + Fluoride varnish (FV)

INTERVENTIONS:
Device: A "simple medical strategy" consisting of silver diamine fluoride (SDF) — Advantage Arrest, Elevate Oral Care LLC., West Palm Beach, FL)
  Other Names: SDF treatment
  Arms: A "simple medical strategy" consisting of SDF
Device: B "typical dental strategy" consisting of atraumatic restorative treatment (ART) with glass ionomer cement + Fluoride varnish (FV) — GC Fuji (for ART) and FluoriMax Advantage Arrest, Elevate Oral Care LLC., West Palm Beach, FL (for FV)
  Other Names: ART + FV treatment
  Arms: A "typical dental strategy" consisting of ART + FV

SUMMARY:
The study is a cluster randomized clinical trial (RCT) to be conducted in 40 (22 originally planned +16 additional) publicly subsidized housing facilities/sites (HUD Section 202) and other low-income housing voucher programs in NE Ohio. The facilities will be randomized to 2 arms: Arm 1 (20 sites) - Participants will receive biannual silver diamine fluoride (SDF) versus Arm 2 (20 sites): Participants will receive atraumatic restorative treatment (ART) with glass ionomer cement (GIC) + biannual fluoride varnish (FV) application. A total of 590 (550 originally planned + 40 additional) participants (Arm 1: 295, Arm 2: 295) will be followed for one year (baseline, 26 weeks, 52 weeks).

The protocol for each arm will address both coronal and root surface tooth decay lesions: Arm 1: The treatment will be bi-annual topical 38% SDF(Advantage Arrest, Elevate Oral Care LLC., West Palm Beach, FL) following manufacturer's instructions and published guidelines; Arm 2: The treatment will be ART will be a modification where the cavity will be restored with high viscosity glass-ionomer cement (GIC) (GC Fuji Automix LC Resin Reinforced Glass Ionomer Restorative, Japan)). Patients will also receive biannual topical fluoride varnish treatments (FluoriMax, Elevate) according to manufacturer's instructions.

DETAILED DESCRIPTION:
Study Design:

A cluster randomized clinical trial (RCT) is planned in 40 (22 originally planned +16 additional) publicly subsidized housing facilities (HUD Section 202) and other low-income housing voucher programs in NE Ohio and will be randomized to 2 arms: Arm 1 (20 sites) - Participants will receive biannual SDF; Arm 2 (20 sites): Participants will receive ART + FV biannual application. All participants will be followed for one year and will receive a dental screening and prophylactic cleaning at all visits.

Study Population and Setting:

The long-term goal is to reduce disparities and improve oral health equity for low-income older adults. The immediate goal is to test interventions to address disparities. Therefore, the population/setting will be low socioeconomic status (SES) adults ≥ 62 years of age in 6 NE Ohio counties (Cuyahoga, Lorain, Summit, Ashtabula, Geauga, and Lake) residing in HUD Section 202 and other publicly subsidized housing facilities. Administrators have provided letters of support confirming the availability of sites and intent to participate. The population is diverse: African American/Black, Caucasian/White including Hispanic/Latino, and Asian. There are 64 HUD housing sites with 3,661 tenant units in the 6 counties. An additional 87 low-income facilities housing elderly are accounted for by regional housing authorities, adding 11,667 units. Therefore, a total of 151 facilities and 15,328 older adults are available.

The sample size goal of 40 (22+16) sites and 590 (550 originally planned + 40 additional) participants will be easily achieved. Medicaid participation among the tenants is 76% among facilities. From a prior study in these facilities it is expected that the mean age is 74 years, 76% female, 51% Caucasian, 45% African-American, 2% Hispanic, and 2% other racial/ethnic groups; 60% of HUD older adults had none/rare dental visits in over 3 years.

Due to COVID-19 restrictions which prevented outside visitors/providers at the housing sites, recruitment will take longer than the anticipated 24 months. Additionally, approximately 40 enrolled individuals did not complete the 26 week visit/second dose of treatment. We therefore increased the total number of enrolled participants by 40 (included in total above). We also added sixteen additional housing facilities to the study to address some delays in recruitment due to the COVID-19 pandemic.

The additional 16 sites will also be randomized to Arm 1 and Arm 2 for a total of 20 sites in each arm

Recruitment of Participants:

Successful strategies from prior studies will be used in recruiting and input will be solicited from the stakeholders. Strategies that will be used are as follows: Service coordinators at all 40 facilities will serve as site liaisons. The study PI/project manager will provide the service coordinators with an introductory letter/flyer containing study information to be given to tenants and to be posted in public areas of the facility. Service coordinators will first arrange an informational meeting (study dentist will give a talk on the interventions as suggested by our stakeholders), and will arrange a second recruitment meeting for study staff to present information regarding the study at scheduled group events (e.g. tenant meetings, health fairs). For planning purposes, service coordinators will have a sign-up sheet for those interested in the sessions. Study staff will schedule those who are interested and meet the inclusion criteria for one-on-one sessions at the housing facility to obtain informed consent and collect baseline survey data. Baseline dental exam and treatment appointments will then be scheduled at each facility according to a designated exam day(s) for each facility, which will occur approximately 1-2 weeks following consent and baseline data collection. Six and twelve month dental exams/treatment and one-on-one interviews for follow-up survey completion for each time point will also occur at the housing facility where participants reside.

Randomization Procedures:

Randomization is at the level of the cluster (housing facility) for logistical efficiency. This will greatly reduce the potential for error that could otherwise occur with people at the same site assigned to different treatments. Furthermore, keeping the same treatment at each site reduces chances of 'contamination' (i.e. participant discussing their treatment with others). Additionally, stratified cluster randomization will be used, i.e. a block (constrained) randomization approach in which balance over treatments is assured for 2 key cluster-level (stratification) variables, namely facility size (>100 versus ≤100 residents), and geographic location (Cuyahoga County vs other). The project statistician will generate the randomization scheme for the 40 housing facilities.

Analytic plan:

Each primary outcome will be compared between the SDF and ART+FV groups. For tooth pain, a 95% confidence interval (CI) based on a t-test for the difference in mean responses (SDF minus ART+FV) will be computed. If this confidence interval lies within the interval (-∞, 8) we may conclude 'non-inferiority' of SDF relative to ART+FV treatment. The confidence interval may secondarily be examined to assess possible superiority of one intervention over the other. For arrest rate, a 95% CI for the difference in rates (based on a z statistic) will be computed. If this confidence interval lies within the interval (-0.09, 1) we may conclude 'non-inferiority' of the SDF relative to ART+FV treatment. As above, possible superiority of one intervention over the other may also be assessed. For other outcomes, computing 95% CI for differences in means (or proportions for binary outcomes) will also be used. These secondary outcomes will be assessed in an exploratory manner for possibly superiority or inferiority based on appropriate margins.

To corroborate initial results, a generalized estimating equations (GEE) approach will be used. For each outcome, a GEE (marginal) model will be fit that includes a treatment indicator and prognostic variables (including sociodemographic variables, medical conditions, and oral health behaviors). Appropriate link functions (e.g., logit link for binary outcomes and identity link for continuous outcomes) will be specified and an exchangeable working correlation matrix used to allow for correlations within site. The arrest outcome will be analyzed as a binary outcome (as described in the sample size section), and secondarily as the number of arrested lesions assuming an appropriate distribution (e.g., negative binomial) and link function (e.g., log link). Robust t tests with correction for a small number of clusters will be used to test for treatment effects and corresponding 95% confidence intervals computed.

Secondarily, the above GEE approach will be extended to analyze the repeated (baseline, 26 and 52 week) measures for each outcome. The models for each outcome will include the same prognostic variables as before, as well as time and a time by treatment interaction. Correlations among the repeated measures will be allowed, e.g., using a first-order autocorrelation structure. If a substantial within-facility correlation is found it would be necessary to incorporate facility as a second cluster levels (within which person - the first cluster level - is nested). Additionally, estimation and testing (via a robust t-test) the interaction term to compare trends over time for the two interventions will also be employed. If the use of two cluster levels is not found to be feasible in the GEE approach, a generalized mixed effects model approach will be considered.

Causal Inference standards: The use of randomization and adjustment in regression models should be sufficient to provide causally interpretable intervention effect estimates; special causal inference techniques such as propensity score or instrumental variable methods often indicated for observational studies, will therefore not be necessary for the data analysis. Biases will be avoided in causal inferences about the intended interventions by using an intent-to-treat approach, in which individuals are analyzed according to randomized groups without regard to (extent of) treatment actually received.

Sensitivity Analyses: Sensitivity of conclusions to model assumptions will be checked as well as methodological decisions such as outcome definition. In particular, for the arrest outcome, the primary analysis is based on a binary indicator of 'complete' arrest of all lesions for an individual. Results will be corroborated from this approach with an alternative approach analyzing number of lesions arrested. For the GEE analyses, planned for all outcomes, sensitivity will be assessed in part by using alternative working covariance structures and alternative sets of predictors. For some outcomes, alternative distributions will be considered; for example, for number of arrested lesions, possible distributions include Poisson, negative binomial, zero-inflated Poisson (ZIP), and zero-inflated negative binomial (ZINB). Sensitivity to assumptions regarding missing data will also be investigated as described further below.

Missing Data. (a) Methods to prevent and monitor missing data: All questionnaires (using tablets) and dental assessment forms (using paper), will be managed in an electronic database (REDCap) by study staff. Weekly quality control checks will be run for outliers, entry errors, missing data, and potential data anomalies. Statistical analyses, summary and missing data reports will be generated by the study biostatistician monthly during the study. (b) Statistical Methods to Handle Missing Data and Account for Statistical Uncertainty Due to Missingness: The primary analyses, which use GEE based on all available observations, assume outcomes are missing completely at random (MCAR). As an initial assessment of missing data patterns, intervention groups (including by relevant subgroups and time point) will be compared with regard to missing outcome rates. A test for a relationship between missingness and outcomes at early time points will evaluate the plausibility of the MCAR assumption. Multiple imputation methods (an established method) will be used to help assure valid inferences. (d) Plans to Record and Report Dropout and Missing Data: The trial data will be managed using REDCap software, currently running at Case Western Reserve University (CWRU). REDCap is a secure web-based application providing an intuitive interface for validated data entry, audit trails for tracking data manipulation and export procedures, and automated export procedures for seamless data downloads to common statistical packages. Missing data reports will be generated weekly from REDCap for timely resolution and reporting purposes. (e) Plans to Examine Sensitivity of Inferences to Missing Data Methods As noted above, multiple imputation will be used to obtain valid inferences in the presence of data that are not missing completely at random. Predictive mean matching with an appropriate prediction model will be used depending on the outcome (e.g. logistic regression for binary outcomes, linear regression for continuous and count outcomes). Alternative imputation models will be used as part of sensitivity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study (1 year)
* Male or female, aged 62 years or older
* Live in a participating older adult housing facility to continue in the clinical trial phase of the study, an individual must:
* Have at least one untreated active root or coronal carious lesion with ICDAS-II (2015) lesion severity code of 3 or greater

Exclusion Criteria:

* Sensitivity to silver or other heavy-metal ions
* Those with ulcerative gingivitis or stomatitis
* Serious life-threatening medical disease

Min Age: 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra S Nelson, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nelson S, Albert JM, Milgrom P. Comparative Effectiveness of Two Nonsurgical Treatments to Reduce Oral Health Disparities From Untreated Tooth Decay in Older Adults: Protocol for a Cluster Randomized Trial. JMIR Res Protoc. 2020 Sep 8;9(9):e17840. doi: 10.2196/17840. PMID 32897236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty (40) low income housing sites were randomized to one of two treatment arms, however, seven (7) were unable to participate due to logistical reasons. Adults aged 62 and older were recruited from the remaining 33 sites in Northeast Ohio from September 2019 - April 2023 to participate in the baseline dental screening (952 completed the screening). The goal was to enroll 590, but only those with active decay (568) were eligible to participate in the clinical trial phase of the study (phase 2).
Pre-assignment Details: Randomization was at the level of the cluster (housing facility)
Units Other Than Participants: Housing Sites
Period: Baseline Visit
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Started | 346; 20 Housing Sites | 222; 20 Housing Sites
Completed | 346; 18 Housing Sites | 222; 15 Housing Sites
Not Completed | 0; 2 Housing Sites | 0; 5 Housing Sites
Period: 26 Week Follow-Up Visit
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Started | 346; 18 Housing Sites | 222; 15 Housing Sites
Completed | 284; 18 Housing Sites | 185; 15 Housing Sites
Not Completed | 62; 0 Housing Sites | 37; 0 Housing Sites
Not completed — Missed due to COVID-19/logistical issues | 51 | 35
Not completed — Withdrawal by Subject | 11 | 2
Period: 52 Week Follow-Up Visit
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Started | 335; 18 Housing Sites (Participants did not have to complete the 26 week follow-up visit to be eligible to complete the 52 week follow-up visit. Therefore, the number of participants starting is higher than the number completing the 26 week follow-up visit.) | 220; 15 Housing Sites (Participants did not have to complete the 26 week follow-up visit to be eligible to complete the 52 week follow-up visit. Therefore, the number of participants starting is higher than the number completing the 26 week follow-up visit.)
Completed | 291; 18 Housing Sites | 195; 15 Housing Sites
Not Completed | 44; 0 Housing Sites | 25; 0 Housing Sites
Not completed — Missed due to COVID-19 or logistical issues | 22 | 13
Not completed — Withdrawal by Subject | 22 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV | Total
Number analyzed (Participants) | 346 | 222 | 568
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.13 (6.95) | 68.85 (6.39) | 69.63 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data was missing for two participants
  Participants
    number analyzed (Participants) | 344 | 222 | 566
    Female | 193 | 98 | 291
    Male | 151 | 124 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 339 | 211 | 550
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 204 | 165 | 369
  White | 122 | 42 | 164
  More than one race | 14 | 8 | 22
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 346 | 222 | 568
Decayed Tooth Surfaces [Mean (Standard Deviation); unit: decayed tooth surfaces] | 5.80 (7.55) | 4.76 (5.81) | 5.39 (6.93)
Tooth Pain and Sensitivity [Mean (Standard Deviation); unit: scores on a scale] — Tooth Pain and Sensitivity were assessed using the PROMIS v.1.0 - Pain Intensity 3a (Modified for Dental). A mean pain intensity score was created for the 3-item scale and ranged from 0-4 (Had no pain - 0, Mild-1, Moderate-2, Severe-3 to Very Severe - 4) and was then collapsed to 0-2 (No pain-0, mild/moderate-1, and severe/very severe-2. Higher score indicate more pain.
  scores on a scale | 0.25 (0.48) | 0.24 (0.49) | 0.24 (0.48)
Geriatric Oral health Related Quality of Life [Mean (Standard Deviation); unit: scores on a scale] — The Geriatric Oral Health Related Quality of Life (GOHRQoL) overall score is created by taking the sum of each of the 12 items, which were collected using a Likert type scale with 3 levels (Always/Often - 1, Sometimes/Seldom - 2, Never - 3). The scores ranged from 12-36 with higher scores indicating better quality of life.
  scores on a scale | 30.03 (4.57) | 29.78 (4.88) | 29.93 (4.69)

OUTCOME MEASURES:

1. Primary Outcome: Caries Arrest Rate
Description: International Caries Detection and Assessment System was the standard used to identify active caries lesions by examination at baseline by calibrated dental hygienists.
  ICDAS examination was then used to assess caries arrest on permanent tooth surfaces with moderate to severe lesions (ICDAS codes 3-6 with activity code 2 (active)) that received SDF or ART + FV treatment baseline. A lesion was considered arrested if, at follow-up, the activity code is 1 (inactive) or the surface is sound (code S). The mean was calculated with standard deviation for both arms.
Time Frame: Baseline to 26 weeks
Population: Analysis was completed for the SDF (279) group and ART + FV group (184).
Measure: Mean (Standard Deviation); unit: surfaces
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 279 | 184
surfaces | 0.75 (0.36) | 0.91 (0.21)

2. Primary Outcome: Caries Arrest Rate
Description: as for outcome 1
Time Frame: Baseline to 52 weeks
Population: Analysis was completed for the SDF (272) group and ART + FV group (187).
Measure: Mean (Standard Deviation); unit: surfaces
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 272 | 187
surfaces | 0.88 (0.25) | 0.92 (0.21)

3. Primary Outcome: Tooth Pain
Description: Tooth Pain and Sensitivity were assessed using the PROMIS v.1.0 - Pain Intensity 3a (Modified for Dental). A mean pain intensity score was created for the 3-item scale and ranged from 0-4 (Had no pain - 0, Mild-1, Moderate-2, Severe-3 to Very Severe - 4) and was then collapsed to 0-2 (No pain-0, mild/moderate-1, and severe/very severe-2. Higher scores indicate more pain.
Time Frame: Baseline to 26 weeks
Population: Analysis was completed for the SDF (284) group and ART + FV group (184) for Pain Scores at 26 weeks.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 284 | 184
scores on a scale | 0.27 (0.50) | 0.21 (0.44)

4. Primary Outcome: Tooth Pain
Description: as for outcome 3
Time Frame: Baseline to 52 weeks
Population: Analysis was completed for the SDF (290) group and ART + FV group (192) for Pain Scores at 52 weeks.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 290 | 192
scores on a scale | 0.21 (0.43) | 0.25 (0.49)

5. Secondary Outcome: Prevention of New Decay
Description: New decay was defined as ICDAS lesion code ≥3 (localized to extensive decay) on one or more surfaces on teeth previously not found at baseline even on surfaces that did not receive the study treatments. ICDAS examination was used to determine the count of newly decayed surfaces on teeth and the mean was calculated.
Time Frame: Baseline and 26 weeks
Population: Analysis for SDF (281) group and ART + FV group (184) for newly decayed surfaces at 26 weeks.
Measure: Mean (Standard Deviation); unit: surfaces
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 281 | 184
surfaces | 0.94 (2.03) | 0.52 (1.46)

6. Secondary Outcome: Prevention of New Decay
Description: as for outcome 5
Time Frame: Baseline to 52 weeks
Population: Analysis for SDF (282) group and ART + FV group (192) for newly decayed surfaces at 52 weeks.
Measure: Mean (Standard Deviation); unit: surfaces
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 282 | 192
surfaces | 0.67 (1.72) | 0.66 (1.71)

7. Secondary Outcome: Oral Health Related Quality of Life
Description: Geriatric Oral Health Related Quality of Life (GOHRQoL) overall score is created by taking the sum of each of the 12 items, which were collected using a Likert type scale with 3 levels (Always/Often - 1, Sometimes/Seldom - 2, Never - 3). The overall scores ranged from 12-36 with higher scores indicating better quality of life. The mean was calculated for the SDF and ART groups.
Time Frame: Baseline to 26 weeks
Population: Analysis for SDF (284) group and ART + FV group (184) for the mean of overall GOHRQoL scores at 26 weeks.
Measure: Mean (Standard Deviation); unit: mean of overall scores on a scale
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 284 | 184
mean of overall scores on a scale | 30.73 (4.33) | 30.45 (4.43)

8. Secondary Outcome: Oral Health Related Quality of Life
Description: as for outcome 7
Time Frame: Baseline to 52 weeks
Population: Analysis for SDF (290) group and ART + FV group (192) for the mean of overall GOHRQoL scores at 52 weeks.
Measure: Mean (Standard Error); unit: mean of overall scores on a scale
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
Number analyzed (Participants) | 290 | 192
mean of overall scores on a scale | 30.44 (4.65) | 30.04 (4.94)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to the 52 week follow-up.
Description: Adverse event information was collected for participants. Adverse events were unrelated to the intervention.
Arm/Group | A "Simple Medical Strategy" Consisting of SDF | A "Typical Dental Strategy" Consisting of ART + FV
All-Cause Mortality (participants affected / at risk) | 14/346 | 8/222
Serious Adverse Events (participants affected / at risk) | 14/346 | 8/222
Other Adverse Events (participants affected / at risk) | 0/346 | 0/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A "Simple Medical Strategy" Consisting of SDF (N=346) | A "Typical Dental Strategy" Consisting of ART + FV (N=222)
Death (General disorders) | 14 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT03916926/Prot_SAP_000.pdf